CLINICAL TRIAL: NCT01629407
Title: A Study of the Rate of Progression of Glaucoma During a Follow-up Period of Two Years
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: MAF/AGN/OPH/GLA/015
Record Dates: First submitted 2012-06-25; First posted 2012-06-27 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2013-06

CONDITIONS: Glaucoma, Open-Angle
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Glaucoma: Patients with glaucoma
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Standard of Care — Patients with glaucoma treated with standard of care at the discretion of the physician. There is no specific treatment required for this study.

SUMMARY:
This is an epidemiological, non-interventional, prospective study to collect data on glaucoma progression in a routine setting. Patients may receive treatment at the discretion of their physician per local standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Glaucoma in one or both eyes

Exclusion Criteria:

* Participation in a glaucoma therapeutic clinical trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with primary open angle glaucoma in one or both eyes
Sampling Method: Non-Probability Sample
Enrollment: 315 (Actual)
Dates: Start 2009-06; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Visual Field | Baseline, 24 Months

SECONDARY OUTCOMES:
Change from Baseline in Intraocular Pressure (IOP) | Baseline, 24 Months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Barcelona, Spain